CLINICAL TRIAL: NCT04350710
Title: Evaluation of Respiratory Mechanics and Lung Recruitment in Patients With SARS-CoV-2 Associated Acute Respiratory Distress Syndrome
Brief Title: Description of Respiratory Mechanics in Patients With SARS-CoV-2 Associated ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2030/31
Record Dates: First submitted 2020-04-09; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Distress Syndrome; COVID
Keywords: COVID; Acute Respiratory Distress Syndrome; SARS CoV-2; Lung recruitability; Respiratory mechanics
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PEEP trial — Measurement of Recruitment-to-Inflation Ratio

SUMMARY:
The aim of this observationnal study is to describe respiratory mechanics and lung recruitement in patients with SARS-CoV-2 Associated Acute Respiratory Distress Syndrome who underwent invasive ventilation on endotracheal tube, admitted to the medical ICU of Angers university hospital . Statics measurements of respiratory system compliance were performed at 2 differents levels of PEEP (15 cmH2O and 5 cmH2O). The recruited volume is computed as the difference between the volume expired from PEEP 15 to 5 cmH2O and the volume predicted by compliance at PEEP 5 cmH2O . The recruitment-to-Inflation (R/I) ratio (i.e. the ratio between the recruited lung compliance and CRS at PEEP 5 cmH2O) is used to assess lung recruitability. A R/I ratio value higher than or equal to 0.5 was used to define highly recruiter patients.

DETAILED DESCRIPTION:
The investigators perform an observational prospective study in patients admitted to medical ICU in Angers University hospital with a confirmed COVID 19 pneumonia and who require invasive ventilation on endotracheal tube. Participants receive initially deep sedation and neuromuscular blockers for 24 hours and are ventilated in volume-controlled mode with a tidal volume of 6 mL/kg of predicted body weight, a constant inspiratory flow of 60 L/minute and a respiratory rate adjusted to maintain pH above 7.35 when possible. A PEEP decremental trial from 15 to 5 cmH2O was performed (15 minutes by step).

Esophageal pressure monitoring and electrical impedance tomography (EIT) are collected if available. Arterial blood gases and respiratory mechanics are measured at the end of each step.

The recruitment-to-Inflation (R/I) ratio (i.e. the ratio between the recruited lung compliance and CRS at PEEP 5 cmH2O) is used to assess lung recruitability. A R/I ratio value higher than or equal to 0.5 is used to define highly recruiter patients.

By the end of the recording time, a low-flow (5 L/min) inflation from PEEP 5 cmH2O (tidal volume = 6ml/kg PBW) is then performed after a prolonged expiration to identify a potential airway closure and the corresponding airway opening pressure (AOP).

Investigators perform these measurements at day 1, day 5 and day 10 from ICU admission if participants still require controlled ventilation.

The investigators also collect clinical data about each participant (past medical history, ICU discharge, hospital discharge, date of death, ventilator acquired pneumonia, thromboembolic event, use of NO, use of ECMO or renal replacement therapy).

ELIGIBILITY:
Inclusion Criteria:

* ARDS criteria according to Berlin classification criteria
* Invasive mechanical ventilation on endotracheal tube
* SARS Cov-2 infection

Exclusion Criteria:

* pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically Ventilated adult patients with COVID-19 Associated ARDS
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-04-20 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment-to Inflation ratio (R/I ratio) | Day 1
  no unit
Recruitment-to Inflation ratio (R/I ratio) | Day 5
  no unit
Recruitment-to Inflation ratio (R/I ratio) | Day 10
  no unit

SECONDARY OUTCOMES:
PaO2/FiO2 (mmHg) | Day 1
  Arterial blood gases
PaO2/FiO2 (mmHg) | Day 5
  Arterial blood gases
PaO2/FiO2 (mmHg) | Day 10
  Arterial blood gases
Lung volume recruited (VRec) | Day 1
  mL
Lung volume recruited (VRec) | Day 5
  mL
Lung volume recruited (VRec) | Day 10
  mL
Plateau pressure (cm H2O) | Day 1
  Obtained by inspiratory pause of 5 seconds
Plateau pressure (cm H2O) | Day 5
  Obtained by inspiratory pause of 5 seconds
Plateau pressure (cm H2O) | Day 10
  Obtained by inspiratory pause of 5 seconds
Oesophagal pressure (cm H2O) | Day 1
Oesophagal pressure (cm H2O) | Day 5
Oesophagal pressure (cm H2O) | Day 10
weight (Kg) | Day 1
weight (Kg) | Day 5
weight (Kg) | Day 10
urine output (mL) | day 1
urine output (mL) | day 5
urine output (mL) | day 10
serum creatinine (Umo/L) | day 1
serum creatinine (Umo/L) | day 5
serum creatinine (Umo/L) | day 10
Mean arterial pressure (mmHg) | day 1
Mean arterial pressure (mmHg) | day 5
Mean arterial pressure (mmHg) | day 10
Peak Pressure (cm H2O) | Day 1
Peak Pressure (cm H2O) | Day 5
Peak Pressure (cm H2O) | Day 10
PEEP total (cm H2O) | Day 1
  Obtained by expiratory pause of 5 seconds
PEEP total (cm H2O) | Day 5
  Obtained by expiratory pause of 5 seconds
PEEP total (cm H2O) | Day 10
  Obtained by expiratory pause of 5 seconds
PEP Set (cm H2O) | Day 1
PEP Set (cm H2O) | Day 5
PEP Set (cm H2O) | Day 10
Height (cm) | Day 1
Airway pening pressure (cm H2O) | day 1
Airway pening pressure (cm H2O) | day 5
Airway pening pressure (cm H2O) | day 10
Expired volume in PEEP setted at 15 cmH2O (mL) | Day 1
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted
Expired volume in PEEP setted at 15 cmH2O (mL) | Day 5
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted
Expired volume in PEEP setted at 15 cmH2O (mL) | Day 10
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted
Expired volume in PEEP setted at 5 cmH2O (mL) | Day 1
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted
Expired volume in PEEP setted at 5 cmH2O (mL) | Day 5
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted
Expired volume in PEEP setted at 5 cmH2O (mL) | Day 10
  respiratory rate decreased to 10 /min, expired tidal volume displayed by the ventilator is noted

CONTACTS AND LOCATIONS:
Overall Officials: François BELONCLE, MCU PH, Principal Investigator — CHU Angers, Médecine intensive réanimation
Locations (1):
- CHU, Angers, France

IPD SHARING:
Plan to Share IPD: No